CLINICAL TRIAL: NCT00030056
Title: Trial of GM-CSF for Alveolar Proteinosis
Brief Title: GM-CSF in Patients With Pulmonary Alveolar Proteinosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: FD-R-002016; FD-R-002016-01
Record Dates: First submitted 2002-01-30; First posted 2002-01-31 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2002-01

CONDITIONS: Pulmonary Alveolar Proteinosis
Keywords: Sargramostim; Injections, Subcutaneous
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

INTERVENTIONS:
Drug: GM-CSF (granulocyte-macrophage colony-stimulating factor, sargramostim)

SUMMARY:
This is a study to determine the efficacy and safety of granulocyte-macrophage colony-stimulating factor (GM-CSF, sargramostim) administered subcutaneously to patients with pulmonary alveolar proteinosis (PAP).

DETAILED DESCRIPTION:
PAP is a rare lung disease characterized by accumulation of surfactant phospholipids and proteins within the lungs. There is no specific pharmacologic therapy for PAP and the current practice of lung lavage under general anesthesia is invasive and has limitations. Although it is unknown if the anti GM-CSF antibody is related to the disease pathogenesis, observations suggest a role for GM-CSF in lung homeostasis as well as in the pathogenesis of PAP.

Patients will receive subcutaneous GM-CSF or placebo once a day and will be followed on an outpatient basis at 2 weeks, and 1, 2, 3, 4, 5 and 6 months after initiation of therapy. Clinical response will determine dosing schedule and will be evaluated by symptom scores, gas exchange data, and chest radiographs.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of primary or idiopathic PAP
* Creatinine no greater than 2 mg/dL
* Bilirubin no greater than 2 mg/dL
* Liver enzymes no greater than 3 times normal
* Women must use an effective method of contraception, be post menopausal, or be surgically sterilized

Exclusion criteria:

* Active respiratory infection
* Active cardiovascular disease (e.g., cardiogenic pulmonary edema)
* Underlying myeloproliferative disorder or leukemia
* Other secondary cause of PAP (e.g., occupational exposure to silica or HIV with PCP)
* At increased risk of side effects from GM-CSF therapy (i.e., rheumatoid arthritis, immune thrombocytopenia, or autoimmune thyroiditis)
* Previous therapy with GM-CSF
* Pregnant or nursing
* Significant renal or liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2001-09; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - National Jewish Medical Center, Denver, Colorado
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The University of Pennsylvania Medical Center, Philadelphia, Pennsylvania